CLINICAL TRIAL: NCT05173922
Title: "Safety in Dementia": An Online Caregiver Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21-4084
Record Dates: First submitted 2021-11-17; First posted 2021-12-30 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Caregivers; Decision Making; Alzheimer Disease; Social Media; Safety; Suicide
MeSH Terms: conditions — Alzheimer Disease; Suicide | interventions — Safety

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety in Dementia (Experimental): Safety in Dementia is an online tool that, in a stepwise fashion, guides a caregiver individual through decisions related to firearm access for a person with dementia. It includes information and a comparison of the options and their risks and benefits. It guides the caregiver through clarification of personal feelings and values and identifying their decision/plan.
  Interventions: Behavioral: Safety in Dementia
- Web control (Active Comparator): The control group will view National Institute on Aging Home Safety Checklist.
  Interventions: Behavioral: Safety in Dementia

INTERVENTIONS:
Behavioral: Safety in Dementia — Safety in Dementia is an online tool that, in a stepwise fashion, guides a caregiver individual through decisions related to firearm access for a person with dementia. It includes information and a comparison of the options and their risks and benefits. It guides the caregiver through clarification of personal feelings and values and identifying their decision/plan. The control group will view national Institute on Aging Home Safety Checklist.

SUMMARY:
In an online randomized trial of Safety in Dementia with national recruitment and longitudinal follow-up, we will recruit informal caregivers of community-dwelling adults with dementia who have firearm access.

DETAILED DESCRIPTION:
Aim 1: To test the efficacy of Safety in Dementia (SiD) on firearm safety decision quality and behaviors, among a national sample of informal caregivers of community-dwelling people with dementia and firearm access (n=500).

Aim 2: To compare varied methods in reaching informal caregivers. Aim 3: To explore stakeholder longitudinal experiences with SiD and firearm-related decisions.

ELIGIBILITY:
Inclusion Criteria:

* Live in United States
* Speak English or Spanish
* Informal caregiver for community swelling person with dementia and firearm access
* Access to the internet

Exclusion Criteria:

* In legal custody or institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Preparation for Decision Making | During baseline assessment (specifically, after receiving randomization allocation), 2 weeks, 2 months, 6 months
  The Preparation for Decision Making Scale assesses perception of how useful a decision aid is in preparing for subsequent decision-making. Scores range from 1-5, calculated from the average of 9 constructs (each ranging from 1, strongly disagree to 5, strongly agree). The scale has high test reliability (0.944) and discriminates significantly between different decision support interventions. In our pilot RCT, participants had a mean score of 3.9 (SD 0.7) after viewing the SiD firearm section.

SECONDARY OUTCOMES:
Change in Decision Self-Efficacy | baseline/pre-intervention, 2 weeks, 2 months, 6 months
  The Decision Self-Efficacy Scale measures confidence in ability to make decisions; transformed scores range from 0 (extremely low) to 100 (extremely high self-efficacy).
Change in Firearm access | baseline/pre-intervention, 2 weeks, 2 months, 6 months
  Firearm access for the person with ADRD will be assessed with scales we have used in prior work, allowing nuanced (but efficient) description of firearm access (on a scale ranging from access to multiple loaded firearms to no access to any firearms). For analysis, we will use binary categorization (any access to 1+ firearm versus no access to any firearms)
Action to reduce firearm access | 2 weeks, 2 months, 6 months
  This will be self-report of taking action to reduce access to one or more firearms (e.g., locking of additional firearm or moving out of the home). The question and categories will allow identification of smaller, albeit important, changes; for analysis we will use binary categorization (any action versus no action).
Firearm injury | baseline/pre-intervention, 2 weeks, 2 months, 6 months
  We will assess injuries or near-miss injuries (e.g., threatening situations) involving the person with ADRD and a firearm. Participants will be asked about any such incidents in the prior year (baseline) or since enrollment (follow-up) and a brief description.
Caregiver burden | 2 weeks
  The short-form Zarit Burden Interview has scores ranging from 0-48, calculated from the sum of 12 items (measured on a 5-point scale from 0, never to 4, nearly always), with scores over 20 indicating high burden.
Positive Aspects of Caregiving | 2 weeks
  The Positive Aspects of Caregiving Scale has scores ranging from 0-36, calculated from the sum of 9 items (measured on a 5-point scale ranging from 0, disagree a lot, to 4, agree a lot, on statements such as feel more useful), with higher scores indicating more positive experiences.
Website analytics | 6 months
  Outcomes obtained from Google analytics will include average minutes spent on Safety in Dementia and specific pages viewed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Betz ME, Portz J, Knoepke C, Ranney ML, Fischer SM, Peterson RA, Johnson RL, Omeragic F, Castaneda M, Greenway E, Matlock D. The Effect of the "Safety in Dementia" Online Tool to Assist Decision Making for Caregivers of Persons With Dementia and Access to Firearms : A Randomized Trial. Ann Intern Med. 2024 Dec;177(12):1630-1640. doi: 10.7326/ANNALS-24-00763. Epub 2024 Oct 22. PMID 39531391
- [Derived] McCarthy V, Portz J, Fischer SM, Greenway E, Johnson RL, Knoepke CE, Matlock DD, Omeragic F, Peterson RA, Ranney ML, Betz ME. A Web-Based Decision Aid for Caregivers of Persons With Dementia With Firearm Access (Safe at Home Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 31;12:e43702. doi: 10.2196/43702. PMID 36719721